CLINICAL TRIAL: NCT04270331
Title: Pain, Agitation, Delirium and Sleep Deprivation Assessment and Management in Intensive Care Units, Thailand: a Before-after Study
Brief Title: Assessment and Management of Pain, Agitation, Delirium and Sleep Deprivation (PADS) in ICU by PADS Protocol, Thailand
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Pitchaya Dilokpattanamongkol, Lecturer, Mahidol University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MURA2020/151
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Pain; Agitation on Recovery From Sedation; Delirium
Keywords: pain; agitation; sedation; delirium; protocol
MeSH Terms: conditions — Pain; Delirium; Psychomotor Agitation

STUDY DESIGN:
Intervention Model Description: A before-after study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A Before group (No Intervention): No protocol assigned
- An After group (Experimental): PADS (pain, agitation, delirium, sleep deprivation assessment and management) protocol assigned
  Interventions: Other: PADS protocol

INTERVENTIONS:
Other: PADS protocol — Assessment and management per PADS protocol
  Arms: An After group

SUMMARY:
The investigators proposed that pain, agitation, delirium and sleep deprivation protocol (PADS) will help improve the patients' outcomes (shortening ICU length of stay, improving ventilator free days, increasing delirium free days) in critically ill patients, a university hospital, Thailand.

DETAILED DESCRIPTION:
Pain is frequently reported in patients admitted to an ICU, with an incidence of up to 50% in medical patients during admission, and increasing up to 80% during standard care procedures. Agitation was also reported in 52% of the patients, typically within 4-9 days after admission. However, there were studies reporting inadequate pain, agitation and delirium assessment and management in real-world clinical practice. The clinical practice guideline for the management of pain, agitation/sedation, delirium, immobility, and sleep disruption in adult patients in the ICU was recently published in 2018 and emphasized routinely monitoring pain, agitation and delirium during ICU admissions. Also, appropriate management of pain and agitation in critically ill patients resulted in reduction in ICU length of stay, hospital length of stay, delirium and mortality. Therefore, structural pain, agitation/sedation, delirium assessment and treatment in the ICUs, Thailand might be necessary.

Since pain, agitation/sedation and delirium protocol has not yet been initiated in ICUs, Thailand, this study is designed as a before-after study in order to assess outcomes by comparing between before and after protocol initiation. The objectives of the study were to document the impact of pain, agitation/sedation, delirium protocol on clinical outcomes of ICU patients admitted to ICUs at Ramathibodi Hospital, a university hospital, Thailand

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years and older)
* Patients admitted to medical or surgical intensive care units

Exclusion Criteria:

* Terminal ill patients, or patients unlikely to survive > 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 509 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
ICU free days | During ICU stay or death or a maximum of 28 days
  Days alive and not stay in ICU

SECONDARY OUTCOMES:
Mechanical ventilator free days | During ICU stay or death or a maximum of 28 days
  Day alive and free of mechanical ventilator
Delirium free days | During ICU stay or death or a maximum of 28 days
  Day alive and free of delirium
Frequency of pain, agitation/sedation, delirium, sleep deprivation assessement | During ICU stay or death or a maximum of 28 days
  Times per patient-days of evaluations during ICU stay
Incidence of in-target pain, agitation/sedation, delirium | During ICU stay or death or a maximum of 28 days
  Times per patient-days of in-target pain, agitation/sedation, delirium during ICU stay
Compliance to PADS protocol | During ICU stay or death or a maximum of 28 days
  Times per patient-days of PADS protocol use by healthcare providers during ICU stay
All-cause hospital mortality | During hospital stay or death or a maximum of 90 days
  Rates of all-cause mortality during hospital stay
Antipsychotics use | During ICU stay or death or a maximum of 28 days
  Type and dose of antipsychotics during ICU stay
Non-benzodiazepines use | During ICU stay or death or a maximum of 28 days
  Type and dose of non-benzodiazepines during ICU stay
Benzodiazepines use | During ICU stay or death or a maximum of 28 days
  Type and dose of non-benzodiazepines during ICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Punchika Luetrakool, MD, Principal Investigator — Ramathibodi hospital, Mahidol university
Locations (1):
- Ramathibodi Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Plan to share individual participant data per request and after 2 years from publications
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Two years after publications
Access Criteria: Per request to researchers via email

REFERENCES:
- [Background] Devlin JW, Skrobik Y, Gelinas C, Needham DM, Slooter AJC, Pandharipande PP, Watson PL, Weinhouse GL, Nunnally ME, Rochwerg B, Balas MC, van den Boogaard M, Bosma KJ, Brummel NE, Chanques G, Denehy L, Drouot X, Fraser GL, Harris JE, Joffe AM, Kho ME, Kress JP, Lanphere JA, McKinley S, Neufeld KJ, Pisani MA, Payen JF, Pun BT, Puntillo KA, Riker RR, Robinson BRH, Shehabi Y, Szumita PM, Winkelman C, Centofanti JE, Price C, Nikayin S, Misak CJ, Flood PD, Kiedrowski K, Alhazzani W. Clinical Practice Guidelines for the Prevention and Management of Pain, Agitation/Sedation, Delirium, Immobility, and Sleep Disruption in Adult Patients in the ICU. Crit Care Med. 2018 Sep;46(9):e825-e873. doi: 10.1097/CCM.0000000000003299. PMID 30113379
- [Background] Barr J, Fraser GL, Puntillo K, Ely EW, Gelinas C, Dasta JF, Davidson JE, Devlin JW, Kress JP, Joffe AM, Coursin DB, Herr DL, Tung A, Robinson BR, Fontaine DK, Ramsay MA, Riker RR, Sessler CN, Pun B, Skrobik Y, Jaeschke R; American College of Critical Care Medicine. Clinical practice guidelines for the management of pain, agitation, and delirium in adult patients in the intensive care unit. Crit Care Med. 2013 Jan;41(1):263-306. doi: 10.1097/CCM.0b013e3182783b72. PMID 23269131
- [Background] Reade MC, Finfer S. Sedation and delirium in the intensive care unit. N Engl J Med. 2014 Jan 30;370(5):444-54. doi: 10.1056/NEJMra1208705. No abstract available. PMID 24476433